CLINICAL TRIAL: NCT00949793
Title: In Vivo Confocal Endomicroscopy of the Brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Carl Zeiss Surgical GmbH (Industry)
Responsible Party: Dr. Gerhard Gaida / Clinical Affairs, Carl Zeiss Surgical GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 002441
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Brain Neoplasms
Keywords: Pathology; Microscopy, Confocal; Microscopy, Fluorescence; Intraoperative Procedures
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Experimental)
  Interventions: Device: Endomicroscope

INTERVENTIONS:
Device: Endomicroscope — Endomicroscopic images are taken at several positions on the tumor.

SUMMARY:
The purpose of the study is to test the feasibility of obtaining interpretable in vivo endomicroscopy images which can be compared with traditional histopathology.

Hypothesis: That a rigid confocal endomicroscope can be used during neurosurgery to provide in vivo histology that enables differentiation of tumour tissue from normal adjacent brain tissue.

DETAILED DESCRIPTION:
Confocal endomicroscopy is a medical imaging modality that allows real-time microscopy to be performed on living tissue in vivo. It is already in clinical use in the fields of gastroenterological endoscopy, laparoscopy, dermatology, gynecology and respiratory medicine. This study represents the first time that confocal endomicroscopy will be evaluated for intraoperative imaging in neurosurgery.

The procedure involves a small endoscope which is placed gently into contact with the brain, providing significant in vivo magnification on a scale similar to that obtained by the pathology laboratory microscope. The captured confocal images will be compared with corresponding histology (tissue that is being removed as part of the indicated neurosurgical procedure). The images will be visually compared among each other and with histology images to detect possible clinically relevant information.

ELIGIBILITY:
Inclusion Criteria:

* All patients with neurosurgical pathology requiring surgery in which tumor resection might be evaluated by using biopsy.

Exclusion Criteria:

* Pregnant women
* Inability to give informed consent
* History of allergy to fluorescein
* Patients on beta-blockers or ACE inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To test of the ability of the surgeon to obtain interpretable images during surgery. | During surgery

SECONDARY OUTCOMES:
To correlate the in vivo endomicroscopy images with traditional histopathology. | one week
To evaluate the usability of the device in the OR environment. | During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nakaji, MD, Principal Investigator — Barrow Neurological Institute, St. Joseph's Hospital and Medical Center
Locations (1):
- Barrow Neurological Institute, St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States